CLINICAL TRIAL: NCT00451178
Title: An Open-label, Randomized, Phase 2 Study of R-CHOP Plus Enzastaurin Versus R-CHOP in the First-Line Treatment of Patients With Intermediate and High-Risk Diffuse Large B-Cell Lymphoma
Brief Title: A Study of Participants With Lymphoma Who Take R-CHOP and Enzastaurin Compared to Participants Who Take R-CHOP Only
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9824; H6Q-MC-S028 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Results first posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — enzastaurin; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- R-CHOP and Enzastaurin (Experimental): R-CHOP includes rituximab plus cyclophosphamide, doxorubicin, vincristine, and prednisone treatment therapies.
  Interventions: Drug: enzastaurin; Drug: rituximab; Drug: cyclophosphamide; Drug: doxorubicin; Drug: vincristine; Drug: prednisone
- R-CHOP (Active Comparator): R-CHOP includes rituximab plus cyclophosphamide, doxorubicin, vincristine, and prednisone treatment therapies.
  Interventions: Drug: rituximab; Drug: cyclophosphamide; Drug: doxorubicin; Drug: vincristine; Drug: prednisone

INTERVENTIONS:
Drug: enzastaurin — 1125 milligrams (mg) then 500 mg, oral, daily, six 21-day cycles or up to 3 years
  Other Names: LY317615
  Arms: R-CHOP and Enzastaurin
Drug: rituximab — 375 milligrams per square meter (mg/m^2), intravenous (IV), Day 1 every 21 days, six 21-day cycles
Drug: cyclophosphamide — 750 mg/m^2, IV, Day 1 every 21 days, six 21-day cycles
Drug: doxorubicin — 50 mg/m^2, IV, Day 1 every 21 days, six 21-day cycles
Drug: vincristine — 1.4 mg/m^2, IV, Day 1 every 21 days, six 21-day cycles
Drug: prednisone — 100 mg, oral, Days 1-5, six 21-day cycles

SUMMARY:
To compare R-CHOP plus enzastaurin versus R-CHOP for progression-free survival (PFS) time measured in participants with intermediate and/or high risk for diffuse large B-cell lymphoma (DLBCL) receiving first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

1. Have a histologically confirmed diagnosis of DLBCL based on the World Health Organization classification (Harris et al. 1999) at the time of original diagnosis. Pathology must be reviewed and confirmed prior to enrollment at the investigational site where the participant is entered. Participants with a prior history of an indolent lymphoma or a histological diagnosis of follicular Grade 3 lymphoma will not be eligible for enrollment.
2. Have received no prior chemotherapy.
3. Have an International Prognostic Index (IPI) score ≥2 at time of original diagnosis.
4. Have a performance status of 0, 1, or 2 on the Eastern Cooperative Oncology group (ECOG) scale.
5. Have adequate organ function as follows:

   * Hepatic: total bilirubin ≤1.5 times the upper limit of normal (x ULN); alanine transaminase (ALT) and aspartate transaminase (AST) ≤1.5 x ULN, (≤5 x ULN, if liver involvement).
   * Renal: serum creatinine ≤1.5 x ULN.
   * Adequate bone marrow reserve: platelets ≥75 x 10^9 per Liter (L), absolute neutrophil count (ANC) ≥1.0 x 10^9 per L, unless there is bone marrow involvement.

   Exclusion Criteria:

   Participants must not:
6. Have received treatment within the last 30 days with a drug (not including enzastaurin) that has not received regulatory approval for any indication at the time of study entry.
7. Are receiving concurrent administration of any other systemic anticancer therapy.
8. Are pregnant or breastfeeding.
9. Are unable to swallow tablets.
10. Are unable to discontinue use of carbamazepine, phenobarbital, and phenytoin at least 14 days prior to study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2007-05; Primary Completion 2012-02 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- United States (25):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beverly Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenbrae, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Springs, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Bend, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Matthews, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Willow Grove, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Everett, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Crosse, Wisconsin

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study included chemotherapy, maintenance therapy (only R-CHOP and enzastaurin treatment arm) and follow-up post treatment for long-term efficacy.
Groups:
- R-CHOP and Enzastaurin: Chemotherapy for up to 6 cycles, 21 days/cycle, with R-CHOP and 500 milligrams (mg) Enzastaurin administered once daily (QD) as four 125-mg tablets, with 1125-mg loading dose [3 tablets, 3 times daily (TID)] on Day 2.
  R-CHOP included:
  * Rituximab: 375 milligrams per square meter (mg/m^2) intravenous (IV) administration on Day 1
  * Cyclophosphamide: 750 mg/m^2 IV administration on Day 1
  * Doxorubicin: 50 mg/m^2 IV administration on Day 1
  * Vincristine: 1.4 mg/m^2 (maximum 2 mg) IV administration on Day 1
  * Prednisone: 100 mg administered orally on Days 1 through 5
  Only this arm eligible for maintenance therapy (500 mg enzastaurin, QD up to 3 years). This included participants (pts) who had complete response (CR), CR-unconfirmed (CRu) and/or were (positron emission tomography) PET-negative. Maintenance therapy allowed, at investigator's discretion, if pts had PR and/or were PET-positive/equivocal, or pts who discontinued therapy before 6 cycles otherwise met response criteria.
- R-CHOP: Chemotherapy for up to 6 cycles, 21 days/cycle, with R-CHOP.
  For each cycle, R-CHOP therapy included:
  * Rituximab: 375 mg/m^2 IV administration on Day 1
  * Cyclophosphamide: 750 mg/m^2 IV administration on Day 1
  * Doxorubicin: 50 mg/m^2 IV administration on Day 1
  * Vincristine: 1.4 mg/m^2 (maximum 2 mg) IV administration on Day 1
  * Prednisone: 100 mg administered orally on Days 1 through 5
Period: Chemotherapy (Up To Six 21-Day Cycles)
Arm/Group | R-CHOP and Enzastaurin | R-CHOP
Started | 58 | 43
Received At Least 1 Dose Study Treatment | 57 | 43
Completed | 40 | 26
Not Completed | 18 | 17
Not completed — Adverse Event | 6 | 6
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Protocol Violation | 2 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Death | 4 | 3
Not completed — Progressive Disease (PD) | 1 | 2
Period: Prior to Maintenance Therapy
Arm/Group | R-CHOP and Enzastaurin | R-CHOP
Started | 40 | 0 (R-CHOP participants were excluded from maintenance therapy and went directly to long-term follow-up.)
Completed | 36 | 0
Not Completed | 4 | 0
Not completed — Physician Decision | 2 | 0
Not completed — PD | 2 | 0
Period: Maintenance Therapy (up to 3 Years)
Arm/Group | R-CHOP and Enzastaurin | R-CHOP
Started | 36 | 0 (R-CHOP participants were excluded from maintenance therapy and went directly to long-term follow-up.)
Completed | 6 | 0
Not Completed | 30 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Death | 1 | 0
Not completed — PD | 10 | 0
Not completed — Continuing Maintenance | 9 | 0
Period: Long-Term Follow-Up (Up to 2 Years)
Arm/Group | R-CHOP and Enzastaurin | R-CHOP
Started | 6 | 26
Completed | 0 | 0
Not Completed | 6 | 26
Not completed — Continuing Follow-Up | 6 | 26

BASELINE CHARACTERISTICS:
Population: Randomized participants who received at least 1 dose of enzastaurin or any drug in the R-CHOP regimen.
Groups:
- R-CHOP and Enzastaurin: Chemotherapy for up to 6 cycles, 21 days/cycle, with R-CHOP and 500 mg Enzastaurin administered QD as four 125-mg tablets, with 1125-mg loading dose (3 tablets, TID) on Day 2.
  R-CHOP included:
  * Rituximab: 375 mg/m^2 IV administration on Day 1
  * Cyclophosphamide: 750 mg/m^2 IV administration on Day 1
  * Doxorubicin: 50 mg/m^2 IV administration on Day 1
  * Vincristine: 1.4 mg/m^2 (maximum 2 mg) IV administration on Day 1
  * Prednisone: 100 mg administered orally on Days 1 through 5
  Only this arm eligible for maintenance therapy (500 mg enzastaurin, QD up to 3 years). This included pts who had CR, CRu and/or were PET-negative. Maintenance therapy allowed, at investigator's discretion, if pts had PR and/or were PET-positive/equivocal, or pts who discontinued therapy before 6 cycles otherwise met response criteria.
- Total: Total of all reporting groups
Arm/Group | R-CHOP and Enzastaurin | R-CHOP | Total
Number analyzed (Participants) | 57 | 43 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (13.55) | 63.3 (12.36) | 63.4 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 34 | 22 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 46 | 39 | 85
  African | 6 | 3 | 9
  Hispanic | 3 | 1 | 4
  East Asian | 2 | 0 | 2
  West Asian | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57 | 43 | 100
International Prognostic Index (IPI) [Mean (Standard Deviation); unit: units on a scale] — IPI: tumor scoring system that divides population into risk groups by assigning 1 point for presence of each variable [age >60; lymphoma Stage III (involvement of lymph node regions, both sides of diaphragm) or Stage IV (disseminated involvement ≥1 extra-lymphatic site with or without associated lymph node involvement); >1 extranodal site; elevated lactate dehydrogenase serum level; and Eastern Cooperative Oncology Group (ECOG) status >1: restrictive but ambulatory; range: 0 (fully active) to 4 (completely disabled)]. Range of IPI scores: 0 (low risk) to 5 (high risk).
  units on a scale | 2.88 (0.803) | 2.84 (0.843) | 2.86 (0.815)

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Time
Description: PFS time is the elapsed time from the date of randomization to the first date of objectively-determined PD or death from any cause. PD was assessed according to International Working Group recommendations (Cheson et al. 1999). PD: Enlarging liver/spleen nodules, new or increased lymph nodes/masses and reappearance of bone marrow infiltrate. For participants not known to have died as of the data cut-off date and who did not have objective PD, PFS was censored at the date of the last objective progression-free disease assessment. For participants who received subsequent anticancer therapy (other than enzastaurin maintenance therapy) prior to objectively determined disease progression or death, PFS was censored at the date of the last objective progression-free disease assessment prior to the date of subsequent therapy.
Time Frame: Randomization to measured PD or death from any cause (up to 55 months)
Population: Randomized participants who received at least 1 dose of enzastaurin or any drug in the R-CHOP regimen who had at least 1 post-baseline efficacy measurement. A total of 34 and 21 participants were censored in the R-CHOP/Enzastaurin and R-CHOP arms, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | R-CHOP and Enzastaurin | R-CHOP
Number analyzed (Participants) | 56 | 42
months | 36.2 [20.2 to NA] — The upper 95% confidence interval was not estimable due to the high rate of censoring. | 22.6 [8.9 to NA] — The upper 95% confidence interval was not estimable due to the high rate of censoring.

2. Secondary Outcome: Percentage of Participants With Complete Response (CR and CRu) and Objective Response [CR, CRu, and Partial Response (PR)] (Overall Response Rate)
Description: CR, CRu, and PR were defined using International Working Group recommendations (Cheson et al. 1999). CR is a complete disappearance of all disease with the exception of nodes. No new lesions. Previously enlarged organs must have regressed and not be palpable. Bone marrow must be negative if positive at baseline. Normalization of markers. CRu does not qualify for CR above, due to a residual nodal mass or an indeterminate bone marrow. PR is a 50% decrease in the sum of the products of diameters for up to 6 identified dominant lesions, including splenic and hepatic nodules from baseline. No new lesions and no increase in the size of liver, spleen or other nodes. The percentage of participants with complete response (CR/CRu) and objective response (Cr/CRu/PR)=(Number of participants whose best overall response was CR/CRu or Cr/CRu/PR)/(Number of participants treated)*100.
Time Frame: Baseline through long-term follow-up (up to 2 years post last dose)
Population: Randomized participants who received at least 1 dose of enzastaurin or any drug in the R-CHOP regimen who had at least 1 post-baseline efficacy measurement.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R-CHOP and Enzastaurin | R-CHOP
Number analyzed (Participants) | 56 | 42
percentage of participants
  Complete Response | 51.8 [38.0 to 65.3] | 42.9 [27.7 to 59.0]
  Objective Response | 83.9 [71.7 to 92.4] | 85.7 [71.5 to 94.6]

3. Secondary Outcome: Percentage of Participants Alive Progression-Free at Year 2 (2-Year PFS Rate)
Description: PD was assessed according to International Working Group recommendations (Cheson et al. 1999). PD: Enlarging liver/spleen nodules, new or increased lymph nodes/masses and reappearance of bone marrow infiltrate. Percentage of participants alive progression-free at Year 2=(Number of participants alive progression free at Year 2)/(Number of participants assessed)*100.
Time Frame: Randomization to measured PD (up to Year 2)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R-CHOP and Enzastaurin | R-CHOP
Number analyzed (Participants) | 56 | 42
percentage of participants | 59 [45 to 73] | 49 [32 to 66]

4. Secondary Outcome: Percentage of Participants With a PET-Negative Scan (PET-Negative Rate)
Description: The percentage of participants with a PET-negative scan=(Number of participants who had a PET-negative scan at Cycle 6)/(Number of participants who had a PET-positive scan at baseline)*100.
Time Frame: Cycle 6 (21 days/cycle)
Population: Randomized participants who received at least 1 dose of enzastaurin or any drug in the R-CHOP regimen who had a PET-positive scan at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R-CHOP and Enzastaurin | R-CHOP
Number analyzed (Participants) | 56 | 39
percentage of participants | 44.6 [31.3 to 58.5] | 41.0 [25.6 to 57.9]

5. Secondary Outcome: Percentage of Participants With Complete Response (CR/CRu) and/or Post-Baseline PET-Negative Scan (Concordance Between Response and PET Scan)
Description: Lesion response was assessed according to International Working Group recommendations (Cheson et al. 1999). CR is a complete disappearance of all disease with the exception of nodes. No new lesions. Previously enlarged organs must have regressed and not be palpable. Bone marrow must be negative if positive at baseline. Normalization of markers. CRu does not qualify for CR above, due to a residual nodal mass or an indeterminate bone marrow. Percentage of participants with CR/CRu and/or PET-negative scan=(Number of participants with complete response and/or PET-negative scan at Cycle 6)/(Number of participants with a PET-positive scan at baseline)*100.
Time Frame: Cycle 6 (21 days/cycle)
Population: Randomized participants who received at least 1 dose of enzastaurin or any drug in the R-CHOP regimen, who had a PET-positive scan at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | R-CHOP and Enzastaurin | R-CHOP
Number analyzed (Participants) | 56 | 39
percentage of participants
  CR/CRu and PET-Negative Post-Baseline | 26.8 | 25.6
  CR/CRu or PET-Negative Post-Baseline | 53.6 | 43.6

6. Secondary Outcome: Event-Free Survival (EFS)
Description: EFS is the elapsed time from the date of randomization to the first date of objectively-determined PD, institution of a new anticancer treatment (other than maintenance therapy), or death from any cause. PD was assessed according to International Working Group recommendations (Cheson et al. 1999). PD: Enlarging liver/spleen nodules, new or increased lymph nodes/masses and reappearance of bone marrow infiltrate. For participants not known to have died as of the data cut-off date, who did not have objectively determined disease progression, and who were not treated with a new anticancer treatment, EFS was censored at the date of the last objectively determined disease-free assessment.
Time Frame: Randomization to measured PD, start of new therapy, or death from any cause (up to 55 months)
Population: Randomized participants who received at least 1 dose of enzastaurin or any drug in the R-CHOP regimen who had at least 1 post-baseline efficacy measurement. A total of 31 and 20 participants were censored in the R-CHOP/Enzastaurin and R-CHOP arms, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | R-CHOP and Enzastaurin | R-CHOP
Number analyzed (Participants) | 56 | 42
months | 36.2 [14.6 to NA] — The upper 95% confidence interval was not estimable due to the high rate of censoring. | 22.6 [8.9 to NA] — The upper 95% confidence interval was not estimable due to the high rate of censoring.

7. Secondary Outcome: Overall Survival (OS)
Description: OS is the elapsed time from the date of study enrollment (baseline) to the date of death from any cause. For participants not known to have died as of the data cutoff date, OS was censored at the last contact date or last date known to be alive, whichever was later.
Time Frame: Baseline to death from any cause (up to 55 months)
Population: Randomized participants who received at least 1 dose of enzastaurin or any drug in the R-CHOP regimen who had at least 1 post-baseline efficacy measurement. A total of 42 and 28 participants were censored in the R-CHOP/Enzastaurin and R-CHOP arms, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | R-CHOP and Enzastaurin | R-CHOP
Number analyzed (Participants) | 56 | 42
months | NA [NA to NA] — The median and 95% confidence interval were not estimable due to the high rate of censoring. | NA [32.3 to NA] — The median and upper 95% confidence interval were not estimable due to the high rate of censoring.

8. Secondary Outcome: Duration of Complete Response (CR or CRu)
Description: Duration of response (DOR) either CR or CRu: Elapsed time from date CR or CRu criteria met to first objectively-determined PD. For responding participants (pts) who died without PD and pts not known to have died as of data cut-off date, who did not have PD, DOR censored at date of last objective progression-free disease assessment. For responding pts who received subsequent systemic anticancer therapy (other than enzastaurin maintenance therapy) prior to PD, DOR was censored at date of last objective progression-free disease assessment prior to subsequent therapy. CR and CRu defined using International Working Group recommendations (Cheson et al. 1999). CR is a complete disappearance of all disease with the exception of nodes. No new lesions. Previously enlarged organs must have regressed and not be palpable. Bone marrow (BM) must be negative if positive at baseline. Normalization of markers. CRu does not qualify for CR above, due to a residual nodal mass or an indeterminate BM.
Time Frame: Time of response to PD (up to 55 months)
Population: Randomized participants who received at least 1 dose of enzastaurin or any drug in the R-CHOP regimen who achieved CR or CRu. A total of 22 and 9 participants were censored in the R-CHOP/Enzastaurin and R-CHOP arms, respectively.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | R-CHOP and Enzastaurin | R-CHOP
Number analyzed (Participants) | 27 | 11
days | NA [813 to NA] — The median and upper 95% confidence interval were not estimable due to the high rate of censoring. | NA [1053 to NA] — The median and upper 95% confidence interval were not estimable due to the high rate of censoring.

9. Secondary Outcome: Participants Who Had Treatment-Emergent Adverse Events (TEAEs) or Died (Evaluate Toxicity and Tolerability of R-CHOP Plus Enzastaurin)
Description: Data presented are the number of participants who experienced at least 1 TEAE, Grade 3 or 4 Common Terminology Criteria for Adverse Events (CTCAE), serious adverse event (SAE), as well as the number of participants who discontinued due to an adverse event (AE) or SAE, who died on therapy, died within 30 days post treatment or within 60 days of first dose. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: First dose through 30 days post study treatment discontinuation (up to 56 months)
Population: Safety Population: Randomized participants who received at least 1 dose of enzastaurin or any drug in the R-CHOP regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | R-CHOP and Enzastaurin | R-CHOP
Number analyzed (Participants) | 57 | 43
Participants
  At Least 1 TEAE | 56 | 43
  At Least 1 Grade 3/4 CTCAE | 50 | 30
  At Least 1 SAE | 35 | 18
  Discontinued due to AE | 10 | 6
  Discontinued due to SAE | 4 | 3
  Died on Therapy (all causes) | 5 | 3
  Died within 30 days post treatment discontinuation | 6 | 3
  Died within 60 days of first dose | 3 | 2

10. Secondary Outcome: PFS of Participants With High or Low Expression of Protein Biomarkers and Correlation of Biomarkers to PFS
Description: Reported is PFS of participants (pts) with high or low biomarker expression levels. PFS: time from randomization to first date of PD/death from any cause. PD assessed according to International Working Group recommendations (Cheson et al. 1999). PD: Enlarging liver/spleen nodules, new/increased lymph node/masses and reappearance of bone marrow infiltrate. For pts who had subsequent anticancer therapy, PFS censored at date of last assessment prior to subsequent therapy. Biomarkers and number of pts censored: EIF4EBP1 Cytoplasm (C) 4,3,7,3; EIF4EBP1 Nucleus (N) 0,2,11,4; EIF4E C 5,2,6,4; EIF4E N 0,0,11,6; HDAC2 N 5,1,5,5; PCREB N 5,3,6,4; PEIF3746 C 4,2,7,4; PEIF3746 N 5,2,6,4; PEIFS209 C 5,2,5,4; PEIFS65 N 7,2,4,4; PEIFT70 C 5,2,6,4; PEIFT70 N 6,4,5,2; P GSK3B C 7,3,4,3; PKCb2 C 4,3,7,3; PS6 C 9,4,1,1; PTEN C 5,2,6,4; PTEN N 3,0,8,6. Correlation of biomarkers with PFS (statistical analyses) reported if high expression groups combined and low expression groups combined each had ≥10 pts.
Time Frame: Randomization to measured PD or death from any cause (up to 55 months)]
Population: Randomized participants who received at least 1 dose of enzastaurin or any drug in the R-CHOP regimen, who had at least 1 post-baseline efficacy measurement and had a reported value for the biomarker measure of interest.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- High Biomarker Expression (R-CHOP and Enzastaurin): Participants with high relative biomarker expression levels who were randomized to R-CHOP and Enzastaurin chemotherapy, up to 6 cycles, 21 days/cycle.
  For each cycle, R-CHOP included:
  * Rituximab: 375 mg/m^2 IV administration on Day 1
  * Cyclophosphamide: 750 mg/m^2 IV administration on Day 1
  * Doxorubicin: 50 mg/m^2 IV administration on Day 1
  * Vincristine: 1.4 mg/m^2 (maximum 2 mg) IV administration on Day 1
  * Prednisone: 100 mg administered orally on Days 1 through 5
  Enzastaurin: 500 mg administered QD as four 125-mg tablets, with 1125-mg loading dose (3 tablets, TID) on Day 2.
  Only R-CHOP and Enzastaurin participants eligible for maintenance therapy (500 mg enzastaurin, QD up to 3 years). This included participants who had CR, CRu and/or were PET-negative. Maintenance therapy allowed, at investigator's discretion, if participants had PR and/or were PET-positive/equivocal, or participants who discontinued therapy before 6 cycles otherwise met response criteria.
- High Biomarker Expression (R-CHOP): Participants with high relative biomarker expression levels who were randomized to R-CHOP chemotherapy, up to 6 cycles, 21 days/cycle.
  For each cycle, R-CHOP included:
  * Rituximab: 375 mg/m^2 IV administration on Day 1
  * Cyclophosphamide: 750 mg/m^2 IV administration on Day 1
  * Doxorubicin: 50 mg/m^2 IV administration on Day 1
  * Vincristine: 1.4 mg/m^2 (maximum 2 mg) IV administration on Day 1
  * Prednisone: 100 mg administered orally on Days 1 through 5
- Low Biomarker Expression (R-CHOP and Enzastaurin): Participants with low relative biomarker expression levels who were randomized to R-CHOP and Enzastaurin chemotherapy, up to 6 cycles, 21 days/cycle.
  For each cycle, R-CHOP included:
  * Rituximab: 375 mg/m^2 IV administration on Day 1
  * Cyclophosphamide: 750 mg/m^2 IV administration on Day 1
  * Doxorubicin: 50 mg/m^2 IV administration on Day 1
  * Vincristine: 1.4 mg/m^2 (maximum 2 mg) IV administration on Day 1
  * Prednisone: 100 mg administered orally on Days 1 through 5
  Enzastaurin: 500 mg administered QD as four 125-mg tablets, with 1125-mg loading dose (3 tablets, TID) on Day 2.
  Only R-CHOP and Enzastaurin participants eligible for maintenance therapy (500 mg enzastaurin, QD up to 3 years). This included participants who had CR, CRu and/or were PET-negative. Maintenance therapy allowed, at investigator's discretion, if participants had PR and/or were PET-positive/equivocal, or participants who discontinued therapy before 6 cycles otherwise met response criteria.
- Low Biomarker Expression (R-CHOP): Participants with low relative biomarker expression levels who were randomized to R-CHOP chemotherapy, up to 6 cycles, 21 days/cycle.
  For each cycle, R-CHOP included:
  * Rituximab: 375 mg/m^2 IV administration on Day 1
  * Cyclophosphamide: 750 mg/m^2 IV administration on Day 1
  * Doxorubicin: 50 mg/m^2 IV administration on Day 1
  * Vincristine: 1.4 mg/m^2 (maximum 2 mg) IV administration on Day 1
  * Prednisone: 100 mg administered orally on Days 1 through 5
Arm/Group | High Biomarker Expression (R-CHOP and Enzastaurin) | High Biomarker Expression (R-CHOP) | Low Biomarker Expression (R-CHOP and Enzastaurin) | Low Biomarker Expression (R-CHOP)
Number analyzed (Participants) | 14 | 10 | 18 | 11
months
  Marker: EIF4EBP1 Cytoplasm: number analyzed (Participants) | 5 | 6 | 13 | 7
  Marker: EIF4EBP1 Cytoplasm | NA [12.9 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | 9.49 [8.2 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | 27.96 [10.9 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | 32.30 [2.4 to 32.3]
  Marker: EIF4EBP1 Nucleus: number analyzed (Participants) | 0 | 2 | 18 | 11
  Marker: EIF4EBP1 Nucleus |  | NA [NA to NA] — The median and the upper and lower 95% confidence interval were not estimable because of the high rate of censoring. | NA [12.9 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | 10.55 [4.5 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring.
  Marker: EIF4E Cytoplasm: number analyzed (Participants) | 9 | 6 | 9 | 6
  Marker: EIF4E Cytoplasm | NA [4.3 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | 21.42 [2.4 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | 27.96 [17.1 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | NA [4.5 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring.
  Marker: EIF4E Nucleus: number analyzed (Participants) | 0 | 1 | 18 | 11
  Marker: EIF4E Nucleus |  | 4.50 [NA to NA] — The upper and lower 95% confidence interval was not estimable because of the high rate of censoring. | NA [12.9 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | 32.30 [8.9 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring.
  Marker: HDAC2 Nucleus: number analyzed (Participants) | 10 | 5 | 7 | 7
  Marker: HDAC2 Nucleus | 27.96 [4.3 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | 10.55 [8.2 to 32.3] | NA [12.9 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | NA [2.4 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring.
  Marker: PCREB Nucleus: number analyzed (Participants) | 11 | 9 | 7 | 4
  Marker: PCREB Nucleus | 24.10 [4.3 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | 10.55 [2.4 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | NA [12.9 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | NA [NA to NA] — The median and the upper and lower 95% confidence interval were not estimable because of the high rate of censoring.
  Marker: PEIF3746 Cytoplasm: number analyzed (Participants) | 7 | 6 | 10 | 6
  Marker: PEIF3746 Cytoplasm | 27.96 [8.2 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | 20.90 [4.5 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | NA [4.3 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | NA [2.4 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring.
  Marker: PEIF3746 Nucleus: number analyzed (Participants) | 8 | 4 | 9 | 8
  Marker: PEIF3746 Nucleus | NA [8.2 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | NA [4.5 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | NA [4.3 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | 32.30 [2.4 to 32.3]
  Marker: PEIFS209 Cytoplasm: number analyzed (Participants) | 7 | 8 | 10 | 5
  Marker: PEIFS209 Cytoplasm | NA [4.3 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | 9.20 [2.4 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | 27.96 [8.2 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | NA [10.5 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring.
  Marker: PEIFS65 Nucleus: number analyzed (Participants) | 11 | 4 | 6 | 8
  Marker: PEIFS65 Nucleus | NA [4.3 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | NA [8.9 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | 27.96 [20.2 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | 32.30 [2.4 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring.
  Marker: PEIFT70 Cytoplasm: number analyzed (Participants) | 6 | 3 | 12 | 9
  Marker: PEIFT70 Cytoplasm | NA [8.2 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | NA [8.9 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | 27.96 [10.9 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | 10.55 [2.4 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring.
  Marker: PEIFT70 Nucleus: number analyzed (Participants) | 10 | 9 | 8 | 3
  Marker: PEIFT70 Nucleus | NA [4.3 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | 32.30 [2.4 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | 27.96 [10.9 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | NA [10.5 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring.
  Marker: P GSK3B Cytoplasm: number analyzed (Participants) | 12 | 8 | 6 | 5
  Marker: P GSK3B Cytoplasm | 27.96 [10.9 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | 21.42 [2.4 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | NA [8.2 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | 9.49 [4.5 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring.
  Marker: PKCb2 Cytoplasm: number analyzed (Participants) | 14 | 7 | 10 | 6
  Marker: PKCb2 Cytoplasm | 27.96 [4.3 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | 10.55 [2.4 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | NA [10.9 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | 20.90 [8.2 to 32.3]
  Marker: PS6 Cytoplasm: number analyzed (Participants) | 14 | 10 | 3 | 2
  Marker: PS6 Cytoplasm | NA [10.9 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | 10.02 [4.5 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | 16.57 [12.9 to 20.2] | NA [2.4 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring.
  Marker: PTEN Cytoplasm: number analyzed (Participants) | 9 | 6 | 9 | 7
  Marker: PTEN Cytoplasm | 27.96 [8.2 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | 21.42 [4.5 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | NA [4.3 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | 9.49 [2.4 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring.
  Marker: PTEN Nucleus: number analyzed (Participants) | 6 | 2 | 12 | 11
  Marker: PTEN Nucleus | 27.96 [10.9 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring. | 6.34 [4.5 to 8.2] | NA [8.2 to NA] — The median and upper 95% confidence interval were not estimable because of the high rate of censoring. | 32.30 [8.9 to NA] — The upper 95% confidence interval was not estimable because of the high rate of censoring.
Statistical Analysis 1: Comparison: High Biomarker Expression (R-CHOP and Enzastaurin) vs High Biomarker Expression (R-CHOP) vs Low Biomarker Expression (R-CHOP); The correlation of biomarker EIF4EBP1 Cytoplasm with PFS; Test type: Superiority or Other; Hazard Ratio (HR) = 0.989, 95% CI 2-sided [0.223 to 4.393] — Hazard ratio comparing PFS of participants with a high expression of EIF4EBP1 Cytoplasm [(R-CHOP and Enzastaurin) and (R-CHOP) combined] versus participants with a low expression of EIF4EBP1 Cytoplasm [(R-CHOP and Enzastaurin) and (R-CHOP) combined]
Statistical Analysis 2: Comparison: High Biomarker Expression (R-CHOP and Enzastaurin) vs High Biomarker Expression (R-CHOP) vs Low Biomarker Expression (R-CHOP and Enzastaurin) vs Low Biomarker Expression (R-CHOP); The correlation of biomarker EIF4E Cytoplasm with PFS; Test type: Superiority or Other; Hazard Ratio (HR) = 1.071, 95% CI 2-sided [0.316 to 3.628] — Hazard ratio comparing PFS of participants with a high expression of EIF4E Cytoplasm [(R-CHOP and Enzastaurin) and (R-CHOP) combined] versus participants with a low expression of EIF4E Cytoplasm [(R-CHOP and Enzastaurin) and (R-CHOP) combined]
Statistical Analysis 3: Comparison: High Biomarker Expression (R-CHOP and Enzastaurin) vs High Biomarker Expression (R-CHOP) vs Low Biomarker Expression (R-CHOP and Enzastaurin) vs Low Biomarker Expression (R-CHOP); The correlation of biomarker HDAC2 Nucleus with PFS; Test type: Superiority or Other; Hazard Ratio (HR) = 1.658, 95% CI 2-sided [0.454 to 6.053] — Hazard ratio comparing PFS of participants with a high expression of HDAC2 Nucleus [(R-CHOP and Enzastaurin) and (R-CHOP) combined] versus participants with a low expression of HDAC2 Nucleus [(R-CHOP and Enzastaurin) and (R-CHOP) combined]
Statistical Analysis 4: Comparison: High Biomarker Expression (R-CHOP and Enzastaurin) vs High Biomarker Expression (R-CHOP) vs Low Biomarker Expression (R-CHOP and Enzastaurin) vs Low Biomarker Expression (R-CHOP); The correlation of biomarker PCREB Nucleus with PFS; Test type: Superiority or Other; Hazard Ratio (HR) = 4.082, 95% CI 2-sided [0.455 to 36.628] — Hazard ratio comparing PFS of participants with a high expression of PCREB Nucleus [(R-CHOP and Enzastaurin) and (R-CHOP) combined] versus participants with a low expression of PCREB Nucleus [(R-CHOP and Enzastaurin) and (R-CHOP) combined]
Statistical Analysis 5: Comparison: High Biomarker Expression (R-CHOP and Enzastaurin) vs High Biomarker Expression (R-CHOP) vs Low Biomarker Expression (R-CHOP and Enzastaurin) vs Low Biomarker Expression (R-CHOP); The correlation of biomarker PEIF3746 Cytoplasm with PFS; Test type: Superiority or Other; Hazard Ratio (HR) = 0.636, 95% CI 2-sided [0.180 to 2.253] — Hazard ratio comparing PFS of participants with a high expression of PEIF3746 Cytoplasm [(R-CHOP and Enzastaurin) and (R-CHOP) combined] versus participants with a low expression of PEIF3746 Cytoplasm [(R-CHOP and Enzastaurin) and (R-CHOP) combined]
Statistical Analysis 6: Comparison: High Biomarker Expression (R-CHOP and Enzastaurin) vs High Biomarker Expression (R-CHOP) vs Low Biomarker Expression (R-CHOP and Enzastaurin) vs Low Biomarker Expression (R-CHOP); The correlation of biomarker PEIF3746 Nucleus with PFS; Test type: Superiority or Other; Hazard Ratio (HR) = 0.362, 95% CI 2-sided [0.083 to 1.576] — Hazard ratio comparing PFS of participants with a high expression of PEIF3746 Nucleus [(R-CHOP and Enzastaurin) and (R-CHOP) combined] versus participants with a low expression of PEIF3746 Nucleus [(R-CHOP and Enzastaurin) and (R-CHOP) combined]
Statistical Analysis 7: Comparison: High Biomarker Expression (R-CHOP and Enzastaurin) vs High Biomarker Expression (R-CHOP) vs Low Biomarker Expression (R-CHOP and Enzastaurin) vs Low Biomarker Expression (R-CHOP); The correlation of biomarker PEIFS209 Cytoplasm with PFS; Test type: Superiority or Other; Hazard Ratio (HR) = 1.522, 95% CI 2-sided [0.473 to 4.901] — Hazard ratio comparing PFS of participants with a high expression of PEIFS209 Cytoplasm [(R-CHOP and Enzastaurin) and (R-CHOP) combined] versus participants with a low expression of PEIFS209 Cytoplasm [(R-CHOP and Enzastaurin) and (R-CHOP) combined]
Statistical Analysis 8: Comparison: High Biomarker Expression (R-CHOP and Enzastaurin) vs High Biomarker Expression (R-CHOP) vs Low Biomarker Expression (R-CHOP and Enzastaurin) vs Low Biomarker Expression (R-CHOP); The correlation of biomarker PEIFS65 Nucleus with PFS; Test type: Superiority or Other; Hazard Ratio (HR) = 0.908, 95% CI 2-sided [0.223 to 3.699] — Hazard ratio comparing PFS of participants with a high expression of PEIFS65 Nucleus [(R-CHOP and Enzastaurin) and (R-CHOP) combined] versus participants with a low expression of PEIFS65 Nucleus [(R-CHOP and Enzastaurin) and (R-CHOP) combined]
Statistical Analysis 9: Comparison: High Biomarker Expression (R-CHOP and Enzastaurin) vs High Biomarker Expression (R-CHOP) vs Low Biomarker Expression (R-CHOP and Enzastaurin) vs Low Biomarker Expression (R-CHOP); The correlation of biomarker PEIFT70 Nucleus with PFS; Test type: Superiority or Other; Hazard Ratio (HR) = 1.843, 95% CI 2-sided [0.432 to 7.867] — Hazard ratio comparing PFS of participants with a high expression of PEIFT70 Nucleus [(R-CHOP and Enzastaurin) and (R-CHOP) combined] versus participants with a low expression of PEIFT70 Nucleus [(R-CHOP and Enzastaurin) and (R-CHOP) combined]
Statistical Analysis 10: Comparison: High Biomarker Expression (R-CHOP and Enzastaurin) vs High Biomarker Expression (R-CHOP) vs Low Biomarker Expression (R-CHOP and Enzastaurin) vs Low Biomarker Expression (R-CHOP); The correlation of biomarker P GSK3B Cytoplasm with PFS; Test type: Superiority or Other; Hazard Ratio (HR) = 0.926, 95% CI 2-sided [0.276 to 3.109] — Hazard ratio comparing PFS of participants with a high expression of P GSK3B Cytoplasm [(R-CHOP and Enzastaurin) and (R-CHOP) combined] versus participants with a low expression of P GSK3B Cytoplasm [(R-CHOP and Enzastaurin) and (R-CHOP) combined]
Statistical Analysis 11: Comparison: High Biomarker Expression (R-CHOP and Enzastaurin) vs High Biomarker Expression (R-CHOP) vs Low Biomarker Expression (R-CHOP and Enzastaurin) vs Low Biomarker Expression (R-CHOP); The correlation of biomarker PKCb2 Cytoplasm with PFS; Test type: Superiority or Other; Hazard Ratio (HR) = 0.985, 95% CI 2-sided [0.320 to 3.033] — Hazard ratio comparing PFS of participants with a high expression of PKCb2 Cytoplasm [(R-CHOP and Enzastaurin) and (R-CHOP) combined] versus participants with a low expression of PKCb2 Cytoplasm [(R-CHOP and Enzastaurin) and (R-CHOP) combined]
Statistical Analysis 12: Comparison: High Biomarker Expression (R-CHOP and Enzastaurin) vs High Biomarker Expression (R-CHOP) vs Low Biomarker Expression (R-CHOP and Enzastaurin) vs Low Biomarker Expression (R-CHOP); The correlation of biomarker PTEN Cytoplasm with PFS; Test type: Superiority or Other; Hazard Ratio (HR) = 0.817, 95% CI 2-sided [0.242 to 2.758] — Hazard ratio comparing PFS of participants with a high expression of PTEN Cytoplasm [(R-CHOP and Enzastaurin) and (R-CHOP) combined] versus participants with a low expression of PTEN Cytoplasm [(R-CHOP and Enzastaurin) and (R-CHOP) combined]

ADVERSE EVENTS:
Arm/Group | R-CHOP and Enzastaurin | R-CHOP
Serious Adverse Events (participants affected / at risk) | 35/57 | 18/43
Other Adverse Events (participants affected / at risk) | 56/57 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-CHOP and Enzastaurin (N=57) | R-CHOP (N=43)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (12) | 3 (5)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (3)
Atrioventricular block (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 4 (4)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Alpha haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 2 (2)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 4 (5)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (3) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | R-CHOP and Enzastaurin (N=57) | R-CHOP (N=43)
Anaemia (Blood and lymphatic system disorders) | 22 (26) | 14 (16)
Leukopenia (Blood and lymphatic system disorders) | 16 (40) | 14 (33)
Lymphopenia (Blood and lymphatic system disorders) | 4 (8) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 33 (77) | 26 (59)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (38) | 18 (38)
Palpitations (Cardiac disorders) | 3 (3) | 2 (2)
Lacrimation increased (Eye disorders) | 6 (8) | 4 (6)
Periorbital oedema (Eye disorders) | 3 (10) | 0 (0)
Vision blurred (Eye disorders) | 5 (8) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 7 (8) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 22 (22) | 18 (25)
Diarrhoea (Gastrointestinal disorders) | 27 (35) | 15 (18)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 4 (4)
Nausea (Gastrointestinal disorders) | 29 (46) | 19 (28)
Stomatitis (Gastrointestinal disorders) | 19 (28) | 10 (13)
Vomiting (Gastrointestinal disorders) | 11 (15) | 3 (3)
Asthenia (General disorders) | 9 (11) | 5 (6)
Chills (General disorders) | 6 (6) | 3 (5)
Fatigue (General disorders) | 30 (37) | 29 (40)
Oedema (General disorders) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 18 (30) | 10 (10)
Pain (General disorders) | 5 (5) | 3 (3)
Pyrexia (General disorders) | 13 (18) | 7 (7)
Candidiasis (Infections and infestations) | 4 (5) | 2 (2)
Oral candidiasis (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Staphylococcal infection (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (11) | 1 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 2/23 (2) | 0/21 (0)
Alanine aminotransferase increased (Investigations) | 3 (4) | 2 (2)
Blood creatinine increased (Investigations) | 4 (7) | 1 (1)
Haemoglobin decreased (Investigations) | 5 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 0 (0)
Platelet count decreased (Investigations) | 3 (4) | 0 (0)
Weight decreased (Investigations) | 9 (9) | 3 (3)
Weight increased (Investigations) | 6 (6) | 1 (1)
White blood cell count decreased (Investigations) | 3 (6) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 14 (17) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 9 (14) | 6 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (6) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (13) | 5 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (12) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 4 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (12) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 17 (20) | 5 (6)
Dysgeusia (Nervous system disorders) | 10 (11) | 4 (4)
Headache (Nervous system disorders) | 9 (12) | 3 (4)
Memory impairment (Nervous system disorders) | 4 (4) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 18 (23) | 8 (9)
Paraesthesia (Nervous system disorders) | 4 (4) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (8) | 6 (6)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2)
Depression (Psychiatric disorders) | 3 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 11 (11) | 9 (10)
Chromaturia (Renal and urinary disorders) | 5 (5) | 0 (0)
Nocturia (Renal and urinary disorders) | 4 (4) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 11 (13)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 26 (26) | 17 (17)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 9 (10) | 5 (5)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 4 (4)
Hypertension (Vascular disorders) | 1 (2) | 3 (3)
Hypotension (Vascular disorders) | 6 (6) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days